CLINICAL TRIAL: NCT01487304
Title: Impact of Professional Societies Recommendations on Practical Use of Hormone Replacement Therapy - Project "WOMAN 2005"
Brief Title: Impact of Professional Societies' Recommendations on Practical Use of Hormone Replacement Therapy
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: KLIM-1937
Record Dates: First submitted 2011-12-05; First posted 2011-12-07 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Menopause; Hormone Replacement Therapy, Post-Menopausal
MeSH Terms: interventions — Hormone Replacement Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Low dose HRT
  Interventions: Drug: Marketed low dose hormone replacement therapy

INTERVENTIONS:
Drug: Marketed low dose hormone replacement therapy — A low dose of marketed HRT products prescribed at the discretion of the treating physician

SUMMARY:
This study is conducted in Europe. The aim of this study is to verify the therapeutic effects of low-dose hormone replacement therapy (HRT) in female patients over adequately long time period in normal clinical practice conditions in the Czech Republic.

ELIGIBILITY:
Inclusion Criteria:

* Post-menopausal

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Post-menopausal women suffering from climacteric symptoms who could benefit a switch from standard therapy to low dose therapy at the discretion of the individual physician
Sampling Method: Probability Sample
Enrollment: 3760 (Actual)
Dates: Start 2005-04; Primary Completion 2006-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Breast tenderness

SECONDARY OUTCOMES:
Patient treatment satisfaction after switch to low dose HRT

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Prague, Czechia

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com